CLINICAL TRIAL: NCT05861921
Title: Clinical Assessment of Single-retainer Lithium Di-silicate Versus Zirconia Resin Bonded Fixed Partial Denture for Replacement of an Anterior Missing Tooth. (Randomized Clinical Trial)
Brief Title: Single-retainer Lithium Di-silicate Versus Zirconia Resin Bonded Bridge for Replacement of an Anterior Missing Tooth.
Acronym: RBFPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Catherine Attef Mounir Nasr, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 5223
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and recruiters will not know the study group to which the next participant will be assigned.
  The trial participants, outcome assessors, and data analysis will be blinded after assignment to interventions.
  Emergency un-blinding: In cases of emergency to decrease or prevent any harms for the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-retainer Lithium Di-silicate Resin Bonded Fixed Partial Denture (Experimental): Intervention will be the delivery of Lithium Di-silicate resin bonded fixed partial denture as final prosthetic restorative material for replacing missing upper anterior tooth.
  Interventions: Other: Single-retainer Lithium Di-silicate Resin Bonded Fixed Partial Denture
- Single-retainer Zirconia Resin Bonded Fixed Partial Denture (Active Comparator): Comparator will be the delivery of Zirconia resin bonded fixed partial denture as final prosthetic restorative material for replacing missing upper anterior tooth.
  Interventions: Other: Single-retainer Lithium Di-silicate Resin Bonded Fixed Partial Denture

INTERVENTIONS:
Other: Single-retainer Lithium Di-silicate Resin Bonded Fixed Partial Denture — Lithium Di-silicate as final restorative material for resin bonded Fixed Partial Denture replacing missing upper anterior tooth.

SUMMARY:
First, Participants in this study will be recruit according to inclusion criteria. Proper examination for the participants (clinically and radiographically). Preparation for abutment tooth for Resin bonded fixed partial denture. Checking and verification for the restoration (trying). Clinical assessment and survival evaluation of the final restoration on delivery and on follow-up every 12 weeks for 12 months.

DETAILED DESCRIPTION:
Examination and diagnosis: Selection and examination of the patients according to inclusion and exclusion criteria. Diagnosis of the patient's chief complaint and teeth that will be involved in this study will be done.

Primary alginate impressions for diagnosis on primary casts and for mounting. The patients will be asked to maintain good oral hygiene measures by using tooth brush twice daily.

Taking a professional pre-operative photo.

Tooth preparation procedure:

1. Preparation of abutment tooth for Resin bonded fixed partial denture according to specific standardized design for both types of final restorations.
2. After tooth preparation, the final impression will be taken for each participant using the intraoral scanner.
3. Fabrication of temporary restoration using composite resin temporary material and cemented using Zinc Oxide eugenol free temporary cement.

Fabrication of final restoration:

Lithium Di-silicate or Zirconia Resin bonded fixed partial denture will be fabricated according to group.

Clinical assessment and survival evaluation of the final restoration on delivery and on follow-up every 12 weeks for 12 months following outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* All subjects are required to be:

  1. From 15-50 years old, to be able to read and sign the informed consent document.
  2. Have no active periodontal or pulpal diseases.
  3. Psychologically and physically able to withstand conventional dental procedures
  4. Maintenance of good oral hygiene.
  5. Able to return for follow-up examinations and evaluation
  6. Patients have missing upper incisor tooth.

Exclusion Criteria:

1. Patient less than 15 or more than 50 years old
2. Patient with active resistant periodontal diseases
3. Patients with poor oral hygiene and uncooperative patients
4. Pregnant women
5. Patients in the growth stage with partially erupted teeth
6. Psychiatric problems or unrealistic expectations
7. Lack of opposing dentition in the area of interest
8. More than one missing tooth in the area of interest

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Clinical assessment in the term of fracture. | 1 year
  United States Public Health Service (USPHS) criteria index in Discrete scores

SECONDARY OUTCOMES:
Clinical assessment in the term of De-bonding. | 1 year
  United States Public Health Service (USPHS) criteria index in Discrete scores
Success and survival rates | 1 year
  Binary as in failed or no failed
Patient satisfaction | 1 year
  Questionnaire in discrete scores

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A. Mounir, Asst. lect., Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No